CLINICAL TRIAL: NCT04595461
Title: Effect of Patient Education Videos on Perioperative Anxiety in Patients Undergoing
Brief Title: Effect of Patient Education Videos on Perioperative Anxiety in Patients Undergoing Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrew Thamboo, Clinical Assistant Professor, Division of Otolaryngology-Head and Neck Surgery, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17-03567
Record Dates: First submitted 2020-09-08; First posted 2020-10-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Standard of care patient education with verbal and written education
  Interventions: Other: Control
- Video Group (Experimental): Patient education supplemented with four short youtube videos regarding chronic rhinosinusitis and endoscopic sinus surgery
  Interventions: Other: Video Education

INTERVENTIONS:
Other: Video Education — Patients receive four short YouTube videos explaining chronic rhinosinusitis and endoscopic sinus surgery
  Arms: Video Group
Other: Control — Standard patient education with verbal and written education
  Arms: Control

SUMMARY:
Chronic rhinosinusitis treatment consists of medical management and surgical intervention. Improving patient education can positively impact perioperative patient experiential outcomes such as anxiety, pain and satisfaction. However, online education materials are often too complex, inaccurate or misleading. The objective of this study was to determine if patient education videos at an appropriate reading level would improve perioperative anxiety in patients undergoing endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* diagnosed with CRS according to Canadian Guidelines
* computer or mobile phone access were included

Exclusion Criteria:

* immunocompromised
* had sinonasal tumours
* history of anxiety, depression, bipolar, or any other mental illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pre-operative Patient Anxiety | 1 hour preoperatively
  Measured with State Trait Anxiety Inventory (range 20-80, higher score shows higher anxiety)
Pre-operative Patient Anxiety | 1 hour preoperatively
  Visual Analogue Scale (1-10, higher score means higher anxiety)

SECONDARY OUTCOMES:
Post-operative Anxiety | 1 week post-operative
  Measured with State Trait Anxiety Inventory (range 20-80, higher score shows higher anxiety)
Post-operative Anxiety | 1 week post-operative
  Visual Analogue Scale (1-10, higher score means higher anxiety)
Post-operative Pain | 1 week post-operative
  Measured via Visual Analogue Scale (1-10, higher score means worse pain)
Post-operative Satisfaction | 1 week post-operative
  Measured via Visual Analogue Scale (1-10, higher score means better satisfaction)
Post-operative medication adherence | 1 week post-operative
  Measured via frequency of nasal irrigation per day

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Thamboo, MD, Principal Investigator — University of British Columbia
Locations (1):
- Saint Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Information can be shared with other researchers on reasonable request